CLINICAL TRIAL: NCT02175901
Title: Prospective, Randomized Controlled Trial Comparing Amoxicillin and Metronidazole Based Bismuth-containing Quadruple Therapy With Amoxicillin and Clarithromycin Based Quadruple Therapy for First-line Helicobacter Pylori Eradication
Brief Title: Amoxicillin/Metronidazole Based Quadruple Therapy for Helicobacter Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Professor of GI Division, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjkls2014006
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Dyspepsia; Peptic Ulcer
Keywords: helicobacter pylori eradication; antibiotic
MeSH Terms: conditions — Dyspepsia; Peptic Ulcer | interventions — Lansoprazole; Proton Pump Inhibitors; Bismuth; Amoxicillin; Anti-Bacterial Agents; Metronidazole; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin/metronidazole (Experimental): Amoxicillin/metronidazole-based quadruple therapy for 14 days: Lansoprazole 30mg bid, Bismuth Potassium Citrate 220mg bid, amoxicillin 1000mg bid, Metronidazole 400mg qid
  Interventions: Drug: Lansoprazole; Drug: Bismuth Potassium Citrate; Drug: Amoxicillin; Drug: Metronidazole
- Amoxicillin/clarithromycin (Active Comparator): Amoxicillin/clarithromycin-based quadruple therapy for 14 days: Lansoprazole 30mg bid, Bismuth Potassium Citrate 220mg bid, Amoxicillin 1000mg bid, Clarithromycin 500mg bid
  Interventions: Drug: Lansoprazole; Drug: Bismuth Potassium Citrate; Drug: Amoxicillin; Drug: Clarithromycin

INTERVENTIONS:
Drug: Lansoprazole — antisecretory drug of each quadruple therapy
  Other Names: proton pump inhibitor
Drug: Bismuth Potassium Citrate — one component of each quadruple therapy
  Other Names: Bismuth
Drug: Amoxicillin — antibiotic of each quadruple therapy
  Other Names: antibiotic
Drug: Metronidazole — antibiotic of the amoxicillin/metronidazole-based quadruple therapy
  Other Names: antibiotic
  Arms: Amoxicillin/metronidazole
Drug: Clarithromycin — antibiotic of the amoxicillin/clarithromycin-based quadruple therapy
  Other Names: antibiotic
  Arms: Amoxicillin/clarithromycin

SUMMARY:
No trial has examined the the efficacy of amoxicillin and metronidazole based quadruple therapy for Helicobacter pylori treatment. The study aims to compare the effectiveness and safety of 14-day amoxicillin-/metronidazole-based quadruple regiment and classical quadruple regiment for Helicobacter pylori eradication.

DETAILED DESCRIPTION:
Helicobacter pylori is the most successful human pathogen infecting an estimated 50% of the global population. It is a common and potentially curable cause of dyspepsia and peptic ulcer disease. Eradication in patients with peptic ulcer or even functional or non-investigated dyspepsia is a cost effective approach.

Most Consensus Conferences and Clinical Guidelines recommend the prescription of a triple therapy including a proton pump inhibitor (PPI) and clarithromycin with either amoxicillin or metronidazole, as first-line treatment. However, the effectiveness of these triple-therapy regimens seems to have diminished over time, largely as a result of emerging resistance of the organism to clarithromycin. Due to the low efficacy achieved with these treatments, they have been deemed as unethical comparators in clinical trials. As antimicrobial resistance becomes more prevalent worldwide, treatment failure rates are likely to continue increasing, suggesting that new regimens for H pylori eradication must be sought.

Bismuth-containing quadruple therapies have been used widely in H. pylori therapy with many permutations of doses and durations and with variable results. Classical bismuth-based quadruple therapy containing a PPI, bismuth, tetracycline and metronidazole has been recommended as the first-line treatment by the Maastricht IV Consensus Conference report and H. pylori Study Group of Chinese Society of Gastroenterology. But this regiment has high rate of side effects because of tetracycline. Standard triple therapy-based, bismuth-containing quadruple Therapy is also an alternative. Though addition bismuth and prolonging treatment duration can overcome H. pylori resistance to clarithromycin, its use as a first-line treatment is limited in areas of high clarithromycin resistance.

Amoxicillin has low resistance rate as well as low percentage of side effects. The combination of amoxicillin and metronidazole in bismuth-containing quadruple therapy may be a better choice, which can avoid clarithromycin resistance and reduce side effects. Therefore, we will do a randomized trial to compare the eradication rate of 14-day amoxicillin and metronidazole based bismuth-containing quadruple therapy with amoxicillin and clarithromycin based quadruple therapy for Helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-investigated/functional dyspepsia or scarred peptic ulcer with indication of H pylori eradication treatment
* Ability and willingness to participate in the study and to sign and give informed consent
* confirmed H pylori infection by at least one of the following methods: C13-urea breath test, histology, rapid urease test or bacterial culture.

Exclusion Criteria:

* patients with peptic ulcer
* previous H. pylori eradication therapy
* Age below 18 years
* major systemic diseases
* previous gastric surgery
* pregnancy or breastfeeding
* allergy to any of the study drugs
* receipt of anti-secretory therapy, antibiotics or bismuth salts 4 weeks prior to inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori | 2 months
  Access eradication rate of H. pylori by intention to treat (ITT) and per-protocol (PP) analysis in each treatment group

SECONDARY OUTCOMES:
Frequency of side effects of each treatment | 2 months
  Score side effects as mild, moderate or severe according to their influence on daily activities

OTHER OUTCOMES:
Minimal inhibitory concentrations (MIC) of antibiotics against each helicobacter pylori clinical isolate | 2 months
  Determine MIC of amoxicillin, clarithromycin, and metronidazole by the twofold agar dilution method.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D., Principal Investigator — RenJi Hospital
Locations (1):
- Shanghai Renji Hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Sun Q, Liang X, Zheng Q, Liu W, Xiao S, Gu W, Lu H. High efficacy of 14-day triple therapy-based, bismuth-containing quadruple therapy for initial Helicobacter pylori eradication. Helicobacter. 2010 Jun;15(3):233-8. doi: 10.1111/j.1523-5378.2010.00758.x. PMID 20557366
- [Background] Lu H, Zhang W, Graham DY. Bismuth-containing quadruple therapy for Helicobacter pylori: lessons from China. Eur J Gastroenterol Hepatol. 2013 Oct;25(10):1134-40. doi: 10.1097/MEG.0b013e3283633b57. PMID 23778309
- [Derived] Zhang W, Chen Q, Liang X, Liu W, Xiao S, Graham DY, Lu H. Bismuth, lansoprazole, amoxicillin and metronidazole or clarithromycin as first-line Helicobacter pylori therapy. Gut. 2015 Nov;64(11):1715-20. doi: 10.1136/gutjnl-2015-309900. Epub 2015 Sep 2. PMID 26338726